CLINICAL TRIAL: NCT00542399
Title: Comparing the Metabolic Control of Once to Twice-daily Insulin Detemir Injections in Children and Adolescence With Type 1 Diabetes Mellitus.
Brief Title: Comparing the Metabolic Control of Once to Twice-daily Insulin Detemir Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rmc004543ctil
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2010-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: levemir; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): once a day
  Interventions: Drug: Levemir (insulin detemir)
- 2 (Experimental): twice a day
  Interventions: Drug: Levemir twice a day

INTERVENTIONS:
Drug: Levemir (insulin detemir) — Levemir once a day
  Arms: 1
Drug: Levemir twice a day — Levemir twice a day
  Arms: 2

SUMMARY:
An open-label, treat to target, intervention study in order to compare the metabolic control of once to twice-daily insulin Detemir injections in children and adolescence with type 1 diabetes mellitus.

All eligible patients will be assigned to receive insulin Detemir once daily before breakfast. Short acting insulin analog, Novorapid, will be used for mealtime insulin. The starting dose of insulin Detemir will be individually determined.Based on self-measured fasting blood glucose levels, insulin doses will be titrated throughout the trial, aiming at pre-breakfast and premeal concentrations of 90-180 mg/dl for subjects aged 6-12 years and 80-130 mg/dl for subjects aged 13-18 years.Patients that after 4 weeks titration phase will not achieve the target blood glucose and up titration of insulin Detemir cannot be done, due to hypoglycemic episodes would be switched to treatment consist of twice daily insulin Detemir. If the target blood glucose are not achieved at the end of the 4 weeks titration phase, but further up titration is possible and patient does not suffer from hypoglycemic episodes, the titration period would be extended and patient would not be switched to treatment with 2 injections of insulin Detemir.When achieving blood glucose targets patient will continue until study end on the maintenance phase.

DETAILED DESCRIPTION:
An open label,treat to target, prospective, intervention study in order to compare the metabolic control of once to twice-daily insulin detemir injections in children and adolescence with type 1 diabetes mellitus.

Study objectives:

1. To assess the efficacy and safety of insulin detemir therapy (once or twice daily) using a treat to target titration protocol for initiating and maintaining therapy in children and adolescents with type 1 diabetes.
2. To evaluate the percentage of patients That will achieve a reduction of 0.5% of HbA1c from baseline to end of study evaluation.
3. To evaluate Incidence of sever, nocturnal, symptomatic and asymptomatic hypoglycemia and glucose excursions of both hyper and hypoglycemia as measured by the area under the curve determined by the CGMS technique.

Treatment plan:

Patients will be assigned to receive insulin detemir once daily before breakfast. Short acting insulin analog , Novorapid, will be used for mealtime insulin. The starting dose of insulin detemir will be individually determined. Based on self-measured fasting blood glucose levels, insulin doses will be titrated throughout the trial, aiming at pre breakfast and premeal concentrations of 90-180 mg/dl for subjects aged 6-12 years and 80-130 mg/dl for subjects aged 13-18 years.

Patients that after 4 weeks titration phase will not achieve the target blood glucose and up titration of insulin Detemir cannot be done, due to hypoglycemic episodes, would be switched to treatment consist of twice daily insulin Detemir.

If the target blood glucose are not achieved at the end of the 4 weeks titration phase, but further up titration is possible and patient does not suffer from hypoglycemic episodes, the titration period would be extended and patient would not be switched to treatment with 2 injections of insulin Detemir.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial related activity
2. Children with type 1 diabetes who have been treated with insulin for at least 12 months prior to the study.
3. Age > 6 years and < 18 years
4. HbA1c > 7.7%
5. Ability and willingness to accept the study conditions and to inject insulin detemir

Exclusion Criteria:

1. Impaired renal function or current renal dialysis.
2. Acute or chronic metabolic acidosis, including diabetic ketoacidosis.
3. Known hypoglycemia unawareness.
4. Known or suspected allergy to trial products.
5. Clinical evidence of active liver disease or impaired hepatic function
6. Participation in another study (with study drug) within the last 3 months prior to this trial.
7. Significant concomitant disease likely to interfere with glucose metabolism
8. Proven eating disorders
9. Malignancy within the last 5 years
10. History of repeated severe hypoglycemia within the last year.
11. Known diabetes retinopathy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
HbA1C | at screening visit, at the middle of the study, at the end of the study and prior to sweetching to twice daily treatment
SBGM | 4-8 times a day
CGMS | 72 hours prior to switching to twice daily treatment and at the end of study
Total daily basal and bolus insulin | will be calculated every visit

SECONDARY OUTCOMES:
documentation of hypoglycemic and hyperglycemic episodes | diary will be collected every visit

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Schneider Children Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Nimri R, Lebenthal Y, Shalitin S, Benzaquen H, Demol S, Phillip M. Metabolic control by insulin detemir in basal-bolus therapy: treat-to-target study in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2013 May;14(3):196-202. doi: 10.1111/pedi.12012. Epub 2013 Jan 4. PMID 23289822